CLINICAL TRIAL: NCT01301976
Title: Nutritional State in Ulcerative Colitis Patients
Brief Title: Nutritional State and Intake Nutrients Assessment in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Other Study IDs: upeclin/HC/FMB-Unesp-49
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Ulcerative Colitis in Remission
Keywords: nutritional state; nutrients intake; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the reason patients are deficient in nutrients intake such as antioxidants vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ulcerative Colitis in remission
* Age > 18 yo

Exclusion Criteria:

* Patients with Ulcerative Colitis in activity
* Those patients with food intake trouble
* Those patients with bowel resected

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ulcerative Colitis in remission
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil